CLINICAL TRIAL: NCT03010709
Title: Multimodality Monitoring Directed Management of Aneurysmal Subarachnoid Haemorrhage
Acronym: MMMSAH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Adel Helmy (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Adel Helmy, Principal Investigator, University of Cambridge
Organization: University of Cambridge (Other)
Other Study IDs: A094232
Record Dates: First submitted 2016-12-14; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Aneurysmal Subarachnoid Haemorrhage; Delayed Ischaemic Neurological Deficit; Induced Hypertension; Partial Brain Tissue Oxygen Tension; Cerebral Microdialysis
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Microdialysates, cerebrospinal fluid and blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Aneurysmal subarachnoid haemorrhage (aSAH) affects up to 10,000 individuals per year in the UK. It accounts for ~5% of strokes, but is responsible for about 25% quality-adjusted life years (QALYs) lost due to stroke. Although early repair of ruptured aneurysms and aggressive postoperative management has improved overall outcomes, it remains a devastating disease with mortality approaching 50%. Survivors are left with neurological injuries that range from subtle cognitive deficit to disabling cerebral infarctions, less than 60% them returning to functional independence.

SAH triggers a series of pathological processes resulting in neuronal damage and consequent neurological deficit termed early brain injury (EBI). Many of the patients who survive the initial bleed, deteriorate days later from delayed ischaemic neurological deficit (DIND), which causes poor outcome or death in up to 30% of patients with SAH. Both of these pathological processes are still poorly understood which limits the number of treatment options.

DIND is treated with blood pressure augmentation to ensure adequate blood flow in the brain. In awake patients, response can be easily and accurately assessed by performing a thorough neurological examination. In patients whose clinical condition demands sedation, intubation and ventilation, assessing response to treatment using the neurological examination is virtually impossible. Multimodality monitoring (MM), primarily microdialysis and brain tissue oxygen tension with catheters inserted into the relevant parts of the brain offer direct assessment of both delivery and utilisation of metabolic substrates at the cellular level. These can be used for early detection of DIND as well as monitoring during blood pressure augmentation. The aim of this study is to establish and validate a clinical protocol for MM derived management of SAH patients, to determine optimal therapies for correcting abnormalities in brain metabolism and explore the relationship between MD and other monitoring modalities.

DETAILED DESCRIPTION:
This is a prospective observational study of patients with poor grade subarachnoid haemorrhage (SAH) caused by a ruptured brain artery aneurysm. The investigators aim to include 100 patients over a 5-year period.

SAH is diagnosed using computer tomography imaging of the brain and the presence of a ruptured aneurysm by means of computer tomography angiogram of the vessels of the head. These two investigations are part of the standard clinical practice for every patient with suspected SAH. Term ''poor grade'' is used for cases of SAH where the patient is unconscious i.e. in a coma as a consequence of this disease and whose clinical condition requires intubation and ventilation (with or without sedation) and thus admission to an intensive care unit. All patients with poor grade SAH admitted to the neurosciences critical care unit will be screened for participation in this study. All poor grade SAH patients are unconscious and thus unable to give informed consent. Therefore, the next-of-kin of all eligible patients will be approached to discuss and consider patient's involvement in the study. If there is no next-of-kin, the treating clinician will be approached as a professional consultee.

Once consent is obtained from next-of-kin, the participants will have the following monitoring instituted:

1. An intracranial access device will be inserted under general anaesthesia with an intracranial pressure (ICP), a Licox partial tension of tissue oxygen (PbtO2) probe and a microdialysis (MD) catheter. Neuromonitors will be inserted into the part of the brain that is supplied by the affected artery. This procedure will be performed on the neurocritical care unit or in theatre if patients are undergoing other operative procedures at the same time. Continuous neuromonitoring will commence. Hourly MD samples will be processed and the leftover samples stored in -80oC for cytokine analysis at a later date. Neuromonitoring will continue for as long as clinically needed and up to 21 days from ictus.
2. All participants will be fitted with a near-infrared spectroscopy monitor (NIRS) . This non-invasive monitor is used to measure tissue haemoglobin concentration and oxygen content continuously and at the bedside.
3. Daily transcranial Doppler (TCD) examinations will be performed at the bedside to assess the caliber of large cerebral arteries. This procedure is used in regular clinical practice to diagnose large vessel spasm which is one of the pathological substrates for delayed cerebral ischaemia (DCI) All participants will have a CT brain perfusion scan between day 3 and day 5 from the initial haemorrhage (ictus) or when clinically needed to assess brain perfusion and possibility of DCI which is part of standard clinical practice. These scans are reviewed and reported by consultant neuroradiologists. If they identify an area (or areas) of reversible ischaemia, researchers will review the position of invasive brain monitors - if these are outside of the area of DCI, additional monitors will be inserted into the identified area of reversible ishaemia. Researchers will then use invasive brain monitors (MD and LiCox) and non-invasive monitoring (NIRS and TCD) to assess the response to standard treatment of cerebral reversible ischaemia which is hypertensive therapy i.e. mean arterial pressure (MAP) augmentation with vasoactive medications.

Repeat CT brain perfusion scan will be performed between days 7 and 10 from the initial haemorrhage or earlier if clinically indicated to assess response to treatment.

Following a 6 month period, researchers will see the patients in outpatient clinic to assess functional outcome. This is part of the patient's standard clinical care as all our patients are offered clinical follow up in this way.

Researchers will collect any biological samples that are available as part of the standard clinical care of the participant and will not subject the participants to any additional procedures. This would consist of:

* left over microdialysate samples that are not used for the standard clinical care of the participant
* daily blood samples if the participant has an arterial line or central venous catheter
* samples of cerebrospinal fluid (CSF) if the participant has an external ventricular drain

ELIGIBILITY:
Inclusion Criteria:

* Aneurysmal Subarachnoid Haemorrhage
* Patient in Neurosciences Critical Care Unit
* Patient likely to survive for at least 24 hours

Exclusion Criteria:

1. Patient unsuitable for microdialysis monitoring

   * bleeding diathesis
   * thrombocytopaenia (platelets < 100 x 10e9 per litre)
2. Non-survivable brain injury i.e. patient not expected to survive more than 24 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with aneurysmal subarachnoid haemorrhage who require intubation and ventilation and admission to the critical care unit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-02; Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Improvement in brain tissue oxygen tension | 10 days
  Brain Tissue Oxygen measured continuously on Neurointensive Care.

SECONDARY OUTCOMES:
Lactate to pyruvate ratio measured by microdialysis | 10 days
  Microdialysis measured LP ratio measured hourly on Neurointensive Care.
Improved functional outcome of patients as measured by the validated and widely used Extended Glasgow Outcome Scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adel Helmy, MBBChir PhD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No